CLINICAL TRIAL: NCT02489474
Title: Association of Genetic Polymorphism and Acute Kidney Injury After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0411
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood obtained from enrolled patients before surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recipients undergoing liver transplantation: Patients undergoing liver transplantation will be included and followed up during the first 72 hours post-liver transplantation in order to confirm the development of acute kidney injury. The patients will be divided into two groups (AKI group vs. non-AKI group) according to the development of acute kidney injury.

SUMMARY:
Some of the liver transplantation recipients experience postoperative acute kidney injury due to various causes including genetic factors. Prevention of postoperative acute kidney injury is essential for postoperative care in liver transplantation recipients. The aim of this study is to investigate the relationship between gene polymorphisms which have been known to be associated with postoperative acute kidney injury, and the occurrence of acute kidney injury after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1) adult patients scheduled for liver transplantation

Exclusion Criteria:

1. Patients on dialysis
2. patients not able to read, or understand the consent form
3. ethnicity, other than asian
4. patients refusal

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury after liver transplantation | 72 hours
  The development of acute kidney injury is defined by the following definition: 50% increase in SCr from the baseline (preoperative value) or a 0.3 mg/dl increase from baseline within 48 h without urine output. The development of acute kidney injury after liver transplantation could correlate with gene polymorphisms, which have been known to be associated with postoperative acute kidney injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea